CLINICAL TRIAL: NCT07143513
Title: Real World Evaluation of Sotorasib Among Chinese Non-Small Cell Lung Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20240175
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Sotorasib; AMG 510
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese Participants Treated with Sotorasib: Adult participants with Kirsten rat sarcoma viral oncogene homolog (KRAS) p.G12C-mutated locally advanced or metastatic non-small cell lung cancer (NSCLC) and previously treated with at least 1 prior systemic therapy that have received sotorasib treatment in either location of BOAO Pilot Zone and Hong Kong SAR will be included in this cohort.
  The duration of evidence collection is from initiation of sotorasib to the end of study period, up to approximately 4 years from the date of the first available sotorasib use in BOAO Pilot Zone of around August 2021.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Participants will have received sotorasib orally daily until disease progression or unacceptable toxicity.
  Other Names: AMG 510

SUMMARY:
The primary objective of this study is to characterize the safety profile of sotorasib.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) as of the index date.
* KRAS p.G12C-mutated locally advanced or metastatic NSCLC.
* Received at least 1 dose of sotorasib.
* Receipt of at least 1 prior systemic therapy before use of sotorasib.
* Obtained ICF, if required.

Exclusion Criteria:

* Documentation of being a non-Chinese ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adult participants with KRAS p.G12C-mutated locally advanced or metastatic NSCLC and previously treated with at least 1 prior systemic therapy that have received sotorasib treatment in either location of BOAO Pilot Zone and Hong Kong SAR.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 4 years
Number of Participants with Adverse Events of Interest, Inclusive of Hepatotoxicity, Interstitial Lung Disease/Pneumonitis, and Renal Toxicity | Up to approximately 4 years
Number of Participants with Treatment-related Adverse Events (AEs) | Up to approximately 4 years
Number of Participants with Treatment-related AEs of Grade 3 or Worse | Up to approximately 4 years
Number of Participants with Serious Treatment-related AEs | Up to approximately 4 years
Number of Participants with Treatment-related AEs Leading to Treatment Discontinuation | Up to approximately 4 years
Number of Participants with Treatment-related AEs Leading to Dose Reduction | Up to approximately 4 years
Number of Participants with Treatment-related AEs Leading to Death | Up to approximately 4 years

SECONDARY OUTCOMES:
Overall Survival (OS) from Initial Date of Sotorasib Use to Date of Death | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- China (3):
  - Boao Evergrande International Hospital, Qionghai, Hainan
  - Boao Super Hospital, Qionghai, Hainan
  - Ruijin-Hainan Hospital Shanghai Jiao Tong University School of Medicine Hainan Boao Research Hospital, Qionghai, Hainan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com